CLINICAL TRIAL: NCT01106599
Title: An Open-label, Phase I, Dose Escalation Study Evaluating the Safety, Tolerability and Pharmacokinetics of GDC-0623 Administered Daily in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study Evaluating the Safety, Tolerability, and Pharmacokinetics of GDC-0623 in Patients With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAP4834g; GO01327 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2010-04-16; First posted 2010-04-20 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Solid Cancers
MeSH Terms: interventions — GDC-0623

ARMS (1):
- A (Experimental)
  Interventions: Drug: GDC-0623

INTERVENTIONS:
Drug: GDC-0623 — Repeating oral dose

SUMMARY:
This is an open-label, multicenter, Phase I dose-escalation study to assess the safety, tolerability, and pharmacokinetics of GDC-0623 in patients with locally advanced or metastatic solid tumors. Patients will be enrolled in one of two stages: a dose-escalation stage (Stage I) followed by an expansion stage (Stage II). Stage I will evaluate the safety, tolerability, and pharmacokinetics of increasing doses of GDC-0623 administered orally on a 21 day on/7-day off dosing schedule.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented, locally advanced or metastatic solid tumors for which standard therapy either does not exist or has proven ineffective or intolerable
* Evaluable disease or disease measurable per RECIST
* Life expectancy >= 12 weeks
* Adequate hematologic and end organ function
* Agreement to use effective form of contraception for the duration of the study
* Consent to provide archival tissue
* For the cohort expansion stage (Stage II): Patients in this cohort must have had no more than four prior systemic therapies for cancer and must have KRAS mutant CRC (Stage II A and B), pancreatic cancer (Stage IIC, or KRAS mutant NSCLC [Stage IID])

Exclusion Criteria:

* History of prior significant toxicity from a MEK pathway inhibitor requiring discontinuation of treatment
* History of parathyroid disorder or history of malignancy-associated hypercalcemia requiring therapy in the last 6 months
* History of retinal vein occlusion (RVO) or predisposing factors to RVO, including uncontrolled hypertension, uncontrolled diabetes, uncontrolled hyperlipidemia, and coagulopathy
* Evidence of visible retinal pathology considered a risk factor for retinal vein thrombosis
* History of glaucoma
* Palliative radiotherapy, experimental therapy, or anti-cancer therapy or major surgical procedure within a specified timeframe prior to first dose of study drug
* Current severe, uncontrolled systemic disease
* History of clinically significant cardiac dysfunction
* History of active gastrointestinal bleeding within 6 months prior to screening
* Clinically significant history of liver disease, current alcohol abuse, or current known active infection with HIV, or hepatitis B or C virus
* Active autoimmune disease
* Uncontrolled ascites
* Pregnancy, lactation, or breastfeeding
* Known brain metastases that are untreated, symptomatic, or require therapy to control symptoms
* For the Exploratory PK Cohorts (Stage IB and Stage IC): Patients who have a history of or ongoing gastro-esophageal reflux disease or peptic ulcer, or who have gastric pathology or history of gastric surgery which could affect absorption of GDC-0623 from the stomach, will be excluded from these cohorts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2010-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Incidence and nature of dose-limiting toxicities (DLTs) | Through study completion or early discontinuation
Incidence, nature, and severity of adverse events and serious adverse events, graded according to NCI CTCAE, v4.0 | Through study completion or early discontinuation
Pharmacokinetic parameters of GDC-0623 (total exposure, maximum and minimum plasma concentrations, time to maximum plasma concentration, elimination half-life) | Through study completion or early discontinuation

SECONDARY OUTCOMES:
Objective response for patients with measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) | Through study completion or early discontinuation
Duration of objective response for patients with measurable disease according to RECIST | Through study completion or early discontinuation
Progression-free survival (PFS) for patients with measurable disease according to RECIST | Through study completion or early discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (4):
- United States (4):
  - Los Angeles, California
  - Sacramento, California
  - Oklahoma City, Oklahoma
  - Nashville, Tennessee